CLINICAL TRIAL: NCT06470880
Title: Circulating Tumour DNA Guided Adaptive BRAF and MEK Inhibitor Therapy
Acronym: DyNAMIc
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: University of Manchester (Other); University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CFTSp175
Record Dates: First submitted 2024-05-13; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Melanoma
Keywords: Adaptive Therapy
MeSH Terms: conditions — Melanoma | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM A: Standard of care (Active Comparator): Continuous dosing of encorafenib 450mg once daily plus binimetinib 45mg twice daily.
  Interventions: Drug: Standard of Care
- ARM B: Adaptive therapy (Experimental): 4 weeks of encorafenib 450mg once daily plus binimetinib 45mg twice daily, followed by adaptive cycles based on ctDNA TAB level
  Interventions: Drug: Adaptive Therapy

INTERVENTIONS:
Drug: Adaptive Therapy — A blood test that measures the amount of tumour DNA circulating in the patient's blood (known as ctDNA) will be conducted every two weeks to check if the cancer cells are still present, and if they are becoming active. The result of this test will allow doctors to monitor the activity of the tumour and judge when to pause and resume encorafenib and binimetinib treatment. This intermittent treatment is called 'adaptive therapy'.
  Arms: ARM B: Adaptive therapy
Drug: Standard of Care — Encorafenib and binimetinib delivered to UK standard of care.
  Arms: ARM A: Standard of care

SUMMARY:
The goal of this clinical trial is to investigate adaptive therapy in late-stage cutaneous melanoma. The main question it aims to answer are:

If the patient having breaks in their treatment allows the less resistant cells to continue to grow, this would result in a tumour with a lower proportion of resistant cells, making the tumour less resistant to the treatment, an increasing the time it takes for the disease to progress?

Participants will

* Receive their allocated treatment regimen until their cancer progresses, they or their doctor withdraw them from the study, or until the study ends, whichever happens first.
* Attend fortnightly visits to hospital.
* Complete EORTC QLQ-C30 and PRO-CTCAE questionnaires, prior to treatment, every 12 weeks and at the point of cancer progression, to assess quality of life.

Researchers will compare the adaptive therapy participant arm with a standard of care arm to answer the research question described above.

DETAILED DESCRIPTION:
Encorafenib and binimetinib given in combination ("the treatment") is a standard of care treatment in the UK for late stage cutaneous melanoma, a skin cancer that starts in the cells that produce skin pigmentation. 'Late stage' means it can't be surgically removed, or has spread. The treatment is taken daily. Resistance to the treatment can develop after about 12-15 months. During this period, the treatment will kill the less resistant cells, meaning the tumour has a greater proportion of cells that are resistant to the treatment.

This study aims to investigate if the patient having breaks in their treatment allows the less resistant cells to continue to grow, this would result in a tumour with a lower proportion of resistant cells, making the tumour as a whole less resistant to the treatment, and increasing the time it takes for the disease to progress. A blood test that measures the amount of tumour DNA circulating in the patient's blood (known as ctDNA) will be conducted every two weeks to check if the cancer cells are still present, and if they are becoming active. The result of this test will allow doctors to monitor the activity of the tumour and judge when to pause and resume treatment. This intermittent treatment is called 'adaptive therapy'. The investigators intend to recruit 40 participants with late stage cutaneous melanoma from NHS hospitals in the UK. Ten will receive the standard, daily treatment, and thirty will receive adaptive therapy. Patients will receive their allocated treatment regimen until their cancer progresses, they or their doctor withdraw them from the study, or until the study ends, whichever happens first. As well as the fortnightly visits to hospital, patients will required to complete EORTC QLQ-C30 and PRO-CTCAE questionnaires in order for their quality of life to be assessed. These will be completed before their treatment starts; every 12 weeks from when they start treatment; and again if their cancer progresses.

ELIGIBILITY:
Inclusion Criteria

At Screening

1. Written and informed consent obtained from participant and agreement of participant to comply with the requirements of the study
2. Histological confirmation of cutaneous melanoma
3. ≥ 18 years of age
4. Stage III un-resectable/ IV disease
5. Measurable disease on CT (thorax, abdomen and pelvis, ± neck if indicated) and/or PET-CT, and CT or MRI (brain) scan (RECIST v1.1)
6. BRAF p.V600E/K/R/D mutation confirmed (exact point mutation must be known)
7. ECOG performance status 0/1/2
8. Prior radiotherapy or radiosurgery must have been completed at least 2 weeks prior to the first dose of study drugs
9. Adequate organ function as defined below:

   i. Haemoglobin ≥ 9 g/dL ii. White blood count ≥ 2 x109/L iii. ANCa ≥ 1.2 x109/L iv. Platelet count ≥ 75 x109/L v. Albumin ≥ 2.5 g/dL vi. Total bilirubinb ≤ 1.5 x ULNa vii. ASTa or ALTa ≤ 3 x ULNa viii. Calculated creatinine clearance ≥ 30ml/min
10. Women of childbearing potential participating in the study (WOCBP see Appendix B for definition) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of study drug.
11. WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drugs plus at least 28 days following last dose of drug (either encorafenib or binimetinib), (see Appendix B).
12. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment plus 90 days (duration of sperm turnover) from last dose of drug (either encorafenib or binimetinib), (see Appendix B).

    At randomisation:
13. Left Ventricular Ejection fraction (LVEF) ≥ 50% or ≥LLNa by ECHO
14. BRAF ctDNA TAB level of ≥15 copies/ml of plasma

Exclusion Criteria

1. Prior systemic targeted BRAF/MEKi therapy for stage IV (metastatic) melanoma (treatment for stage III allowed as long as RFS ≥26 weeks following discontinuation of drugs)
2. BRAF wild-type malignant melanoma
3. Metastasis to the brain or leptomeninges
4. Any contraindication to treatment with encorafenib or binimetinib as per the local Summary of Product Characteristics
5. Hypersensitivity to the active substance or to any of the excipients of encorafenib or binimetinib
6. Current use of a prohibited medication as described in Section 8.9
7. History of another malignancy. Exception: Patients who have been disease-free for 3 years, (i.e. patients with second malignancies that are indolent or definitively treated at least 3 years ago), curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS); stage 1, grade I endometrial carcinoma, or patients with a history of completely resected non-melanoma skin cancer. No additional therapy should be required whilst the patient is on study
8. Any serious or unstable pre-existing medical conditions (aside from malignancy exceptions specified above), psychiatric disorders, or other conditions that could interfere with the patient's safety, obtaining informed consent, or compliance with study procedures
9. Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection
10. Patients with rare hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption
11. Child Pugh B or C liver disease
12. Coronary syndromes (including myocardial infarction within 6 months or unstable angina)
13. A history or evidence of current ≥ Class II congestive heart failure as defined by the NYHA guidelines with an ejection fraction of <50% (see appendix C)
14. Treatment refractory hypertension defined as a blood pressure of systolic >150 mmHg and/or diastolic >95 mm Hg on >3 occasions which cannot be controlled by anti-hypertensive therapy
15. Uncorrectable electrolyte abnormalities > CTCAE v5 Grade 1 (e.g. hypokalaemia, hypomagnesaemia, hypocalcaemia), long QT syndrome (baseline 1 QTC interval ≥ 480msec) or taking medicinal products known to prolong the QT interval
16. A history or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR) including presence of predisposing factors to RVO or CSR (e.g., uncontrolled glaucoma or ocular hypertension, uncontrolled hypertension, uncontrolled diabetes mellitus, or a history of hyperviscosity or hypercoagulability syndromes)
17. Females who are pregnant or breast-feeding and are not able to stop breast-feeding prior to first dose of study drugs (see section 7.5)
18. Prisoners or patients who are involuntarily incarcerated
19. Patients who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
To measure tumour response to re-introduction of encorafenib plus binimetinib following the first "drug off " period. | 3 years (Longitudinally throughout the study)
  Specific measure: Maximal reduction in percentage ctDNA mutant BRAF copies/ml of plasma from baseline 2 TAB level upon restart of E+B following first drug off period.

SECONDARY OUTCOMES:
To measure the thresholds of percentage reduction in TAB level in ctDNA as a measure of response to stop drugs and the percentage increase in TAB as a decision to restart drugs. | 3 years (Longitudinally throughout the study)
  Specific measure: ctDNA mutant BRAF copies/ml of plasma
To measure maximal response (complete response (CR)/partial response (PR)/stable disease (SD)/progressive disease (PD)) to therapy in Arm A vs. Arm B | Randomisation until RECIST progression/clinical deterioration (estimated 12 months)
  Specific measure: Maximal radiological response (complete response (CR)/partial response (PR)/stable disease (SD)/progressive disease (PD)) using RECIST v1.1 criteria
To measure progression free survival (PFS) in Arm A vs. Arm B | 3 years (Continuously throughout the study)
  Specific measure: Percentage of participants who have experienced disease progression or death. PFS defined as time from randomisation to radiological (RECIST v1.1 and in Arm B defined as radiological progression whilst on targeted therapy unless stopped due to toxicity/choice) progression
To measure time to clinical deterioration in Arm A vs. Arm B. | 3 years (Continuously throughout the study)
  Specific measure:Time to clinical deterioration. Defined as either the point of radiological progression (defined as per RECIST v1.1) or in participants treated beyond radiological progression, at the time of clinically determined deterioration defined at the discretion of the treating clinician, specifically due to progression of the underlying cancer
To measure overall survival in Arm A vs. Arm B | 3 years (Continuously throughout the study)
  Specific measure: Overall survival (OS) defined as time from randomisation until death from any cause
To measure melanoma specific overall survival in Arm A vs. Arm B | 3 years (Continuously throughout the study)
  Specific measure: Overall survival (OS) defined as time from randomisation until death from melanoma
To measure number of adaptive therapy cycles completed by participants on Arm B | 3 years (Longitudinally throughout the study)
  Specific measure: Number of adaptive therapy cycles completed
To measure median duration of adaptive therapy cycles completed by participants on Arm B | 3 years (Longitudinally throughout the study)
  Specific measure: Median duration of adaptive therapy cycles
To measure whether ctDNA result can be provided within 5 working days from sample receipt into NBC | 3 years (Longitudinally throughout the study)
  Specific measure: Percentage of ctDNA results reported within 5 days from sample receipt into NBC
To measure quality of life in Arm A vs. Arm B | 3 years (Longitudinally throughout the study)
  Specific measure: EORTC QLQ-C30 (standardised tool, scored as outlined by EORTC)
To measure quality of life in Arm A vs. Arm B | 3 years (Longitudinally throughout the study)
  Specific measure: PRO-CTCAE (standardised tool, scored as outlined by NIH)
To measure toxicity (all grade adverse events) in Arm A vs. Arm B | 3 years (Continuously throughout the study)
  Specific measure: Adverse Events and Serious Adverse Events defined by CTCAE version 5

IPD SHARING:
Plan to Share IPD: No
Grouped, anonymised data will be made available after the study has ended.